CLINICAL TRIAL: NCT06079905
Title: Palliative NonOperative Management (PNOM) in Selected Elderly With a Limited Life Expectancy Who Sustained a Proximal Femoral Fracture (PNOM-Implementation); an Implementation Study
Brief Title: Palliative NonOperative Management in Selected Elderly With a Limited Life Expectancy Who Sustained a Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dr. E.M.M. (Esther) Van Lieshout PhD MSc (Other)
Responsible Party: Sponsor-Investigator, Dr. E.M.M. (Esther) Van Lieshout PhD MSc, Associate professor Trauma Surgery, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2023-0270
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail elderly with limited life expectancy that fracture a hip: Frail elderly with limited life expectancy that fracture a hip
  Interventions: Other: Nonoperative treatment; Other: Operative treatment

INTERVENTIONS:
Other: Nonoperative treatment — Nonoperative treatment
Other: Operative treatment — Operative treatment

SUMMARY:
The primary and main aim of this study is to implement PNOM in all hospitals in the Netherlands, so that the selected frail elderly people with a limited life expectancy who fracture a hip receive the care that best meets their needs in the last phase of life. The treatment decision is made through shared decision-making.

Study design: This project is an implementation project, consisting of 4 phases. The main design is a multicenter prospective cohort study.

Study population: The target population are frail (institutionalized) elderly who have a limited life expectancy and fracture their proximal femur. The population that meets this criterion are persons of 70 years or older, who either live in a nursing home or receive a similar level of care at home or in another type institution, and have at least one of the following characteristics: 1) are malnourished (cachexia or a Body Mass Index, BMI, of <18.5 kg/m2); 2) mobility issues with increased risk of falling pretrauma (Functional Ambulation Category, FAC, 2 or less); or 3) have severe comorbidities (American Society of Anesthesiologists, ASA, class 4 or 5).

Methods:

Phases 3 and 4: Installation of a local implementation team, followed by PNOM protocol implementation. Data collection for patients eligible for PNOM by automated data extraction from the national hip fracture audit.

DETAILED DESCRIPTION:
Rationale: A hip fracture in a select group of frail elderly people can indicate an approaching end of life. These patients do not benefit from an operative treatment that aims to restore mobility. The FRAIL-HIP study has shown that palliative non-operative management (PNOM) can be a good alternative for this group. By shared decision making between the patient/family and the medical specialists involved, surgery or PNOM was chosen. Half of the patients opted for PNOM. Quality of life was valued equally by patients in both groups. The majority of the next of kin in both groups rated the quality of dying as very good. The aim of this project is to implement PNOM in all Dutch hospitals as part of shared decision-making in a select group of frail patients with a hip fracture.

Objective(s): The primary and main aim of this study is to implement PNOM in all hospitals in the Netherlands, so that the selected frail elderly people with a limited life expectancy who fracture a hip receive the care that best meets their needs in the last phase of life. The treatment decision is made through shared decision-making. Secondary aims, needed to achieve the main aim, are: 1) to enriching the draft version of the PNOM protocol, and test results of the PNOM protocol draft; 2) to develop educational modules for the curriculum of residents Surgery and Orthopedics; 3) to create awareness and a sense of urgency for PNOM implementation in this select group of patients by organizing PNOM informational sessions during annual conferences of the scientific associations involved; 4) to improve the PNOM protocol on a smaller scale based on implementation of the PNOM protocol in selected hospitals across the country; and 5) to facilitate the scaling up of the implementation of the PNOM protocol to all hospitals in the Netherlands that treat the targeted patient group Study design: This project is an implementation project, consisting of 4 phases. The main design is a multicenter prospective cohort study.

Study population: The target population are frail (institutionalized) elderly who have a limited life expectancy and fracture their proximal femur. The population that meets this criterion are persons of 70 years or older, who either live in a nursing home or receive a similar level of care at home or in another type institution, and have at least one of the following characteristics: 1) are malnourished (cachexia or a Body Mass Index, BMI, of <18.5 kg/m2); 2) mobility issues with increased risk of falling pretrauma (Functional Ambulation Category, FAC, 2 or less); or 3) have severe comorbidities (American Society of Anesthesiologists, ASA, class 4 or 5).

Methods: This study will use mixed methods in the different phases of the study.

Phase 1: interviews with health care professionals and a panel from an elderly person's organization (i.e., patient representatives).

Phase 2: Interviews with patient representatives, development of educational modules for hospitals and residents (Orthopedic) Surgery, and design of a website.

Phases 3 and 4: Installation of a local implementation team, followed by PNOM protocol implementation. Data collection for patients eligible for PNOM by automated data extraction from the national hip fracture audit.

In phase 3, the following additional data will be collected: 1) interviews with health care professionals in the hospital before and at 6 months after start of PNOM implementation; and 2) interviews with patients/proxy/next of kin about their view on the implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Frail institutionalized elderly person (i.e., 70 years or older, living in a nursing home or receiving similar care at the same level while living elsewhere pretrauma, who either are malnourished (cachexia or BMI<18.5 kg/m2), or had mobility issues (FAC 2 or less), or have an ASA class of 4 or 5)
2. Acute proximal femoral fracture, confirmed on X-ray or CT-scan

Exclusion Criteria:

- None

Ages: 70 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: frail (institutionalized) elderly who have a limited life expectancy and fracture their proximal femur
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Nonoperative treatment | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zeelenberg ML, Oosterwijk PC, Willems HC, Gosens T, Den Hartog D, Joosse P, Loggers SAI, Nijdam TM, Pel-Littel RE, Polinder S, Schuijt HJ, Wijnen HH, Van der Velde D, Van Lieshout EMM, Verhofstad MHJ; NOM-Implementation study group. Shared decision-making for non-operative management versus operative management of hip fractures in selected frail older adults with a limited life expectancy: a protocol for a nationwide implementation study. BMJ Open. 2024 Apr 17;14(4):e083429. doi: 10.1136/bmjopen-2023-083429. PMID 38631829